CLINICAL TRIAL: NCT01768507
Title: The Effects of the Dietary Supplement Trans-resveratrol on Heme Oxygenase-1 (HO-1) and Sirtuins Expression in PBMCs in Healthy Male Subjects: A Pilot Study.
Brief Title: Reresveratrol Administered to Healthy Male Subjects
Acronym: REVAHS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Daniel Doberer (Other)
Responsible Party: Sponsor-Investigator, Daniel Doberer, Investigator, Medical University of Vienna
Organization: Medical University of Vienna (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: ClinPharm 754
Record Dates: First submitted 2013-01-13; First posted 2013-01-15 (Estimated); Last update posted 2016-09-15 (Estimated); Status verified 2016-09

CONDITIONS: Healthy Subjects; Heme Oxygenase
MeSH Terms: interventions — Resveratrol

ARMS (2):
- Placebo (Placebo Comparator): no medication
  Interventions: Dietary Supplement: Resveratrol
- Resveratrol (Experimental): Trans-resveratrol (Resveratrol - Terraternal®): 5 g (10 capsules) as single oral dose on day 1 of the investigation period.
  Interventions: Dietary Supplement: Resveratrol

INTERVENTIONS:
Dietary Supplement: Resveratrol — 5 g (10 capsules) as single oral dose on day 1

SUMMARY:
Heme oxygenase 1 (HO-1) serves as a protective gene. The aim of this clinical trial is to evaluate the HO-1 stimulation of resveratrol in healthy humans.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent prior to any study-mandated procedure.
* Male patient aged between 18 and 45 years (inclusive) at screening.
* No clinically significant findings on the physical examination at screening.
* Body mass index (BMI) between 18 and 28 kg/m2 (inclusive) at screening.
* Non-smoker (for at least 1 month)
* Hematology, clinical chemistry, and urinalysis test results not deviating from the normal range to a clinically relevant extent at screening.
* Negative results from urine drug screen at screening.
* Ability to communicate well with the investigator, in the local language, and to understand and comply with the requirements of the study.

Exclusion Criteria:

* Known hypersensitivity to resveratrol or any excipients of the resveratrol formulation.
* Treatment with any investigational drug within 3 weeks prior to screening.
* History or clinical evidence of alcoholism or drug abuse within the 3-year period prior to screening.
* History or clinical evidence of any disease and/or existence of any surgical or medical condition, which might interfere with the absorption, distribution, metabolism or excretion of resveratrol.
* Smoker
* Previous treatment with any prescribed or OTC medications (including herbal medicines such as St John's Wort) within 2 weeks prior to screening.
* Regularly intake of resveratrol rich food
* Positive results from the hepatitis serology at screening.
* Positive results from the HIV serology at screening.
* Presumed non-compliance.
* Legal incapacity or limited legal capacity at screening.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2011-03; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
The maximal HO-1 and sirtuin mRNA expression in PBMCs | 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Austria